CLINICAL TRIAL: NCT02327156
Title: The Effect of a Low-dose Dexmedetomidine as an Adjuvant to Levobupivacaine in Patients Undergoing Vitreoretinal Surgery Under Sub-Tenon's Anesthesia
Brief Title: Dexmedetomidine as an Adjuvant for Sub-Tenon's Anesthesia
Acronym: Precedex
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Magrabi Eye & Ear Hospital (Other)
Responsible Party: Principal Investigator, Ashraf M Ghali, SENIOR CONSULTANT, Magrabi Eye & Ear Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: MEEC-IRB-2014-1
Record Dates: First submitted 2014-12-18; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Vitreoretinal Surgery Under Sub-Tenon's Anesthesia
Keywords: Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group L (No Intervention): receive 4 mL of levobupivacaine 0.75% plus hyaluronidase 15 IU diluted with 1mL normal saline
- group LD (Active Comparator): 4 mL of levobupivacaine 0.75% plus hyaluronidase 15 IU and dexmedetomidine 20 μg diluted with 1mL normal saline
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — adding dexmedetomidine to the local anesthetic
  Other Names: Precedex, 200 μg per 2 mL; Hospira, USA
  Arms: group LD

SUMMARY:
The investigator evaluated the motor and sensory block durations and the postoperative analgesic effects of adding dexmedetomidine to levobupivacaine for sub-Tenon's anesthesia in patients undergoing vitreoretinal surgery. Motor and sensory block durations were considered as a primary endpoint.

DETAILED DESCRIPTION:
Background: The investigator evaluated the motor and sensory block durations and the postoperative analgesic effects of adding dexmedetomidine to levobupivacaine for sub-Tenon's anesthesia in patients undergoing vitreoretinal surgery. Motor and sensory block durations were considered as a primary endpoint.

Methods: The investigator investigated 60 patients subjected to vitreoretinal surgery under sub-Tenon's anesthesia. The patients were randomly divided equally into 1 of 2 groups conferring to the local anesthesia (LA) solution used to receive either 4 mL of levobupivacaine 0.75% plus hyaluronidase 15 IU diluted with 1mL normal saline (group L) or 4 mL of levobupivacaine 0.75% plus hyaluronidase 15 IU and dexmedetomidine 20 μg diluted with 1mL normal saline (group LD). The total volume of the LA solution used was 5 mL. Motor block (akinesia) and sensory block durations were evaluated until the return of normal motor and sensory function. The sedation level was assessed during the surgery period and 24 hours postoperatively together with the degree of postoperative pain and the efficiency of postoperative analgesia. The sleep quality of the first postoperative night was assessed using the Consensus Sleep Diary (CSD).

ELIGIBILITY:
inclusion criteria:

* satisfactory akinesia
* predictable surgical time to be less than 3 hours were inclusion criteria for this study

Exclusion Criteria:

* incorporated patients younger than 18 years,
* patients with a single eye,
* history of sleep apnea,
* severe cardiac disease, and
* drug abuse or
* if there was any contraindication to LA.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
the motor and sensory block durations | participants will be followed for the duration of hospital stay, an expected average of 24 hours
  expected to be extended in group LD

SECONDARY OUTCOMES:
sleep quality of the 1st postoperative night | 24 hours
  improved the sleep quality